CLINICAL TRIAL: NCT06078072
Title: Biomaterials and Mesenchymal Stem/Stromal Cells in the Treatment of Knee Articular Surface Lesions
Status: Completed | Type: Observational
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Sponsor
Other Study IDs: University Medical Centre
Record Dates: First submitted 2023-08-02; First posted 2023-10-11 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-10

CONDITIONS: Knee Injuries; Cartilage Injury; Osteochondral Defect
Keywords: Biomaterials; Mesenchymal stem/stromal cells; Bone marrow aspirate; Cartilage; Osteochondral lesion; Knee
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Biomaterials augmented with mesenchymal stem/stromal cells — Combined single-step procedure of treating knee articular surface lesions with biomaterials (scaffolds) and mesenchymal stem cells (filtered bone marrow aspirate concentrate)

SUMMARY:
The goal of this observational study is to evaluate the combined single-step approach with biomaterials and mesenchymal stem/stromal cells in the treatment of knee articular surface lesions. The clinical analysis of the treatment outcomes, regarding postoperative improvements and safety, is going to be accompanied with laboratory analysis of the intraoperatively applied cellular products.

The main hypothesis are: (1) such combined single-step procedure significantly improves patients' functioning and quality of life; (2) this therapeutic approach is safe; (3) cellular parameters of the applied filtered bone marrow aspirate (fBMA) impact treatment outcomes, among other potential predictors.

Researchers will compare subjective (questionnaire) and objective (clinical examination) status of patients before and after the operation, record any potential complications and perform regression analysis to assess the influence of potential predictors on postoperative improvements.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* patients treated with combined single-step procedure (scaffold and fBMA) for knee articular surface lesions, between January 2013 and December 2020
* symptomatic knee articular surface lesions (International cartilage repair society (ICRS) grades 3-4, size ≥ 1.5 cm2) unresponsive to conservative treatment,
* only mild concomitant osteoarthritis (Kellgren-Lawrence grades 1-2)

Exclusion Criteria:

* patients that refuse to participate in the study
* non responders to the invitation to answer PROMs at the follow-up
* associated medical conditions (inflammatory, metabolic, neoplastic, etc.) that could directly handicap the musculoskeletal system or indirectly impact the quality of life

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 100-150 adult patients (age:18-65) with knee articular surface lesions (size ≥ 1.5 cm2, ICRS grades 3-4) surgically treated with the combined single-step approach (scaffold and fBMA) between January 2013 and December 2020.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Knee injury and Osteoarthritis Outcome Score (KOOS) subscale Pain postoperative improvement | At least 24 months after the operation
  Knee injury and Osteoarthritis Outcome Score (KOOS) assesses patients' pain (9 items), other symptoms (7 items), function in daily living (17 items), function in sport and recreation (5 items), and knee related quality of life (4 items). Scores range from 0 to 100 with a score 0 being the worst score and 100 indicating no impairment.
  KOOS subscale Pain postoperative improvement will be calculated as difference between preoperative and postoperative scores at the final follow up.
  Paired Student t test will be applied to compare preoperative and postoperative values of KOOS subscale Pain.

SECONDARY OUTCOMES:
Knee injury and Osteoarthritis Outcome Score (KOOS) subscales postoperative improvements | At least 24 months after the operation
  Originally published in 1998, the Knee injury and Osteoarthritis Outcome Score (KOOS) assesses patient pain (9 items), other symptoms (7 items), function in daily living (17 items), function in sport and recreation (5 items), and knee related quality of life (4 items). Scores range from 0 to 100 with a score 0 being the worst score and 100 indicating no impairment.
  KOOS subscales postoperative improvements will be calculated as differences between preoperative and postoperative scores at the final follow up. As secondary outcome measures will be calculated all KOOS subscales improvements, beside KOOS subscale Pain, which is determined as the primary outcome measure.
  Paired Student t test will be applied to compare preoperative and postoperative values of all KOOS subscales.
Complications (SAE and GF) | Recording until the final follow up (minimum 24 months after the operation)
  Serious adverse events (SAE) are defined as any hospitalization or revision surgery (arthrofibrosis, synovitis, infection, hardware problem, pulmonary embolism, etc.), while graft failures (GF) as revision surgery to the lesion or confirmed indication for it. SAE will be further classified as related (arthrofibrosis, synovitis, graft hypertrophy/delamination, etc.) or unrelated (hardware removal, meniscus or ligament injuries, new cartilage lesions, pulmonary embolism, etc.) to the graft.
Cellular parameters of intraoperatively applied filtered Bone Marrow Aspirate (fBMA) | Finsihed in 14 days after the procedure
  Samples for cell counting (100 µl), fibroblast colony forming units (CFU-F) assay (1-2 ml) and flow cytometry (1-2 ml) will be taken before and after BMA processing with filter-based separation device. The total nucleated cell (TNC) count will be determined by counting white blood cells with hematology analyzer COULTER® Ac·T diff2™ (Beckman Coulter, Fullerton, CA, USA). MSCs content will be estimated with flow cytometry (FACSCalibur, BD Biosciences, San Jose, CA, USA) by determining CD271+ and CD45-cells, and concomitant assessment of their viability using 7-amino-actinomycin D (7-AAD) dye. Also, the CFU-F assay, which is a functional assay for measuring the frequency of MSCs with the colony forming abilities, will be performed. Briefly, cells will be seeded at least in duplicates into well culture plates and cultured in standard conditions: 37 °C, 5% CO2. After 14 days, colonies containing ≥ 50 fibroblastic cells will be manually counted under the stereomicroscope.
Tegner Activity Scale (TAS) postoperative improvement | At least 24 months after the operation
  Tegner Activity Scale (TAS) is a one-item score that graded activity based on work and sports activities on a 11-level scale from 0 to 10. Zero represents disability because of the knee problems and 10 represents national or international level soccer.
  TAS postoperative improvement will be calculated as difference between preoperative and postoperative scores at the final follow up.
  Paired Student t test will be applied to compare preoperative and postoperative values of TAS.
European Quality of Life 5 Dimensions 3 Level (EQ-5D-3L) postoperative improvement | At least 24 months after the operation
  EQ-5D-3L descriptive system consists of 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression . Each dimension has 3 levels: no problems, some problems, and extreme problems. The respondent is asked to indicate his or her health state by ticking the box that marks the most appropriate level of problems in each dimension. A unique health state can be described according to the responses to the 5 questions. Health states defined in this way may be converted into a single summary index by applying a formula that attaches values to each of the levels in each dimension. States can be converted to a single value where 1 is equivalent to full health and 0 to a state equivalent to death.
  EQ-5D-3L postoperative improvement will be calculated as difference between preoperative and postoperative scores at the final follow up.
  Paired Student t test will be applied to compare preoperative and postoperative values of EQ-5D-3L .
EuroQol Visual Analogue Scale (EQ-VAS) postoperative improvement | At least 24 months after the operation
  EQ-VAS records the patient's self-rated health on a vertical visual analogue scale from 0 to 100, where 0 represents the worst health state imaginable and 100 represents the best health state imaginable.
  EQ-VAS postoperative improvement will be calculated as difference between preoperative and postoperative scores at the final follow up.
  Paired Student t test will be applied to compare preoperative and postoperative values of EQ-VAS5.
Potential predictors (patients' demographics, medical history, joint and lesions' characteristics, surgical and cellular parameters) of the clinical outcomes (KOOS subscales, EQ-5D-3L, EQ-VAS, TAS) | At the time of statistical analysis
  Regression models will be used to assess the influence of proposed predictors (patients' demographics, medical history, joint and lesions' characteristics, surgical and cellular parameters) on the postoperative improvements in clinical outcome measures (KOOS subscales, EQ-5D-3L, EQ-VAS, TAS). Statistical analysis will be performed with SPSS (version 25.0; IBM, Chicago, IL, USA).

CONTACTS AND LOCATIONS:
Overall Officials: Matic Kolar, MD, Principal Investigator — University Medical Centre Ljubljana
Locations (1):
- University medical centre Ljubljana, Ljubljana, Slovenia

REFERENCES:
- [Derived] Kolar M, Veber M, Girandon L, Drobnic M. A Biomimetic Osteochondral Scaffold Augmented With Filtered Bone Marrow Aspirate for the Treatment of Joint Surface Lesions in the Knee. Am J Sports Med. 2024 Jun;52(7):1826-1833. doi: 10.1177/03635465241247788. Epub 2024 May 20. PMID 38767159